CLINICAL TRIAL: NCT04422080
Title: Retrospective Observational Study of Posterior Keratometry Measured by IOLMaster 700 in Patients With Keratoconus
Brief Title: Retrospective Observational Study of Posterior Keratometry Measured
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0338
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Keratoconus
Keywords: Ophthalmology; Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Keratoconus patient: Patient with keratoconus disease diagnosed on videotopography
- Healthy patient: Patient consulting for keratoconus screening with no keratoconus on videotopography

SUMMARY:
Keratoconus is a progressive bilateral disease leading to an apical stromal thinning and an irregular astigmatism by a steepening of the cornea, causing visual impairment. The causes are not yet well known, but it seems to be linked to several comorbidities. Keratoconus is a rare and for a long-time asymptomatic condition and its diagnosis needs meticulous screening for the early stages. Detecting it as soon as possible is a goal as it could lead to earlier avoiding of contributing factors such as eye rubbing and earlier treatment if needed.

The gold standard for keratoconus screening and staging is computerized videotography. It gives information about anterior and posterior corneal bulging, steepening, and thinning. It can be completed by anterior segment optical coherence tomography, which can show corneal scarring. Since recently, some biometry devices can give some information about the posterior corneal keratometry trough swept source optical coherence tomography measures. The measurement of the total corneal power instead of an extrapolation lead to better precision in refractive results after cataract surgery in some cases. It also helped to increase our knowledge about posterior corneal astigmatism. In normal eyes, average posterior corneal astigmatism is 0.37 diopters and against the rule in 91 percent of eyes. There is a correlation between the magnitude of anterior and posterior astigmatism.

In keratoconus eyes, several studies have shown that there is an alignment between axes of the anterior and posterior corneal astigmatism. These studies have been performed on computerized videotopography devices.

The goal of this study was to confirm or deny previous observations about posterior astigmatism in keratoconus eyes, and to assess if the rotation of axis between anterior and posterior astigmatism measured by IOL Master 700® can be a good sign for detection of early stages and fruste keratoconus.

ELIGIBILITY:
Inclusion criteria:

- Keratoconus diagnosed on videotopography

Exclusion criteria:

- loss of sight due to another condition than keratoconus, corneal scarring leading to lack or mistaken data, corneal graft, non-keratoconus related corneal ectasia such as post Laser in Situ Keratomileusis (LASIK) ectasia or keratoglobus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: included all patients having a specialized cornea consultation, in which keratoconus was diagnosed or suspected from November 2018 to May 2020 in the department of Ophthalmology, University Hospital Gui de Chauliac in Montpellier (France),
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Posterior keratometry | 1 day
  Posterior cylinder and axis measured on biometry

SECONDARY OUTCOMES:
Total keratometry | 1 day
  Total corneal power (cylinder and axis) measured on biometrycompleted by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud : MUYL CIPOLLINA, Internship of ophthalmology, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC